CLINICAL TRIAL: NCT04754711
Title: Interest of Nutritional Care of Children With Sickle Cell Disease on Bone Mineral Density and Body Composition
Acronym: NUTRIDREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRO-2020-17
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease; Osteoporosis; Osteopenia
Keywords: Sickle cell disease; Osteoporosis; Osteopenia; bone mineral density; Nutrition; body composition; Oral nutritional supplement
MeSH Terms: conditions — Anemia, Sickle Cell; Osteoporosis; Bone Diseases, Metabolic | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Randomization of patients included in 2 groups
  * Group 1: receiving an oral nutritional supplement to increase calorie intake by around 20%
  * Group 2: "controls" receiving normal calorie intake without oral nutritional supplement Randomization will take into account age, gender and severity of disease in order to create two homogenous groups
  Monitoring by biphotonic absorptiometry, dietetic, clinical and biological
  Creation of a sero-type blood bank for the 2 groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with oral nutritional supplement (Experimental): Group 1: receiving an oral nutritional supplement to increase calorie intake by around 20%
  Interventions: Dietary Supplement: Oral Nutritional Supplement
- Control group (No Intervention): Group 2: "controls" receiving normal calorie intake without oral nutritional supplement

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Supplement — We will propose to the patients of group 1 several different oral nutritional supplements according to taste, and consistency of each child in order to optimize observance. Each of those different oral nutritional supplements will be adapted to the nutritional survey and the age of children without exceeding recommended intake of proteins, carbohydrates, lipids and micronutrients. Those patients will consume the Oral Nutritional Supplement during 12 months.
  Arms: Group with oral nutritional supplement

SUMMARY:
This study is design to assess the effects of an increase in nutritional intake on the bone mineral density of children with sickle cell disease, for 12 months.

DETAILED DESCRIPTION:
* Sickle cell disease is the most common inherited disease of the red blood cell
* During sickle cell disease, the decrease in Bone Mineral Density (BMD) in children is very common: 19 and 56% depending on the studies
* children with sickle cell disease have an increase in resting energy expenditure of 15-20%
* children with sickle cell disease have a significant decrease in muscle mass
* there are no specific nutritional recommendations for sickle cell disease in children

Our main purpose is to assess the effects of an increase in nutritional intake on the bone mineral density of children with sickle cell disease, for 12 months

Our secondary objectives are :

1. / Evaluate the effects of an increase in nutritional intake on: body composition, height and weight growth, frequency of complications of sickle cell disease, school absenteeism, cardiac function, cerebral vasculopathy, biological parameters follow-up, and the relationship with the treatment started
2. / Creation of a sero-type blood bank for future research

ELIGIBILITY:
Inclusion Criteria:

* Following genotypes of sickle cell disease: SS, SC, SE, Sbeta + or Sbeta0
* Ages 3 to 16 years old

Exclusion Criteria:

* Overweight at the start of the study
* Child for whom one of the 2 parents refuses his child's participation in the study

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
The change in the mean Bone Mineral Density of the two randomized groups | Baseline
  The change in the mean Bone Mineral Density of the two randomized groups will be measured by biphotonic absorptiometry (in g/cm2).
The change in the mean Bone Mineral Density of the two randomized groups | Month 12
  The change in the mean Bone Mineral Density of the two randomized groups will be measured by biphotonic absorptiometry (in g/cm2).

SECONDARY OUTCOMES:
Change in body composition | Baseline
  Change in body composition expressed by lean mass (%), fat mass (%), bone mass, by region of the body and overall
Change in body composition | Month 12
  Change in body composition expressed by lean mass (%), fat mass (%), bone mass, by region of the body and overall
Rate of participants with Change of Height | Baseline
  Height-to-age growth in cm and percentile according WHO
Rate of participants with Change of Height | Month 12
  Height-to-age growth in cm and percentile according WHO
Rate of participants with Change of Weight | Baseline
  Weight-to-age growth in kg and percentile according WHO
Rate of participants with Change of Weight | Month 12
  Weight-to-age growth in kg and percentile according WHO
Assessment of school absenteeism | Baseline
  Questionnaire of school absenteeism
Assessment of school absenteeism | Month 3
  Questionnaire of school absenteeism
Assessment of school absenteeism | Month 6
  Questionnaire of school absenteeism
Assessment of school absenteeism | Month 9
  Questionnaire of school absenteeism
Assessment of school absenteeism | Month 12
  Questionnaire of school absenteeism
The frequency of complications of sickle cell disease | Month 12
  Complications such as chronic pain, acute anemia, infections
The presence or not of impaired cardiac function and / or cardiac anatomy related to sickle cell disease | Baseline
  The presence or not of impaired cardiac function and / or cardiac anatomy related to sickle cell disease determined by echocardiography
The presence or not of impaired cardiac function and / or cardiac anatomy related to sickle cell disease | Month 12
  The presence or not of impaired cardiac function and / or cardiac anatomy related to sickle cell disease determined by echocardiography
The presence or not of cerebral vasculopathy | Baseline
  The presence or not of a cerebral vasculopathy sought by transcranial Doppler
The presence or not of cerebral vasculopathy | Month 12
  The presence or not of a cerebral vasculopathy sought by transcranial Doppler
Value change of F-S-C hemoglobin | Baseline
Value change of F-S-C hemoglobin | Month 12
Value change of serum Lactate DeHydrogenase value | Baseline
Value change of serum Lactate DeHydrogenase value | Month 12
Value change of serum iron and ferritin | Baseline
Value change of serum iron and ferritin | Month 12
Value change of serum folate | Baseline
Value change of serum folate | Month 12
Value change of serum C Reactive Protein value | Baseline
Value change of serum C Reactive Protein value | Month 12
Value change of serum 25-OH vitamin D | Baseline
Value change of serum 25-OH vitamin D | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Georges DIMITROV, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: Yes
After the completion and publication of the original study, anonymised data will be made available upon reasonable request to the corresponding author.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the publication of the original research

REFERENCES:
- [Background] Schnog JB, Duits AJ, Muskiet FA, ten Cate H, Rojer RA, Brandjes DP. Sickle cell disease; a general overview. Neth J Med. 2004 Nov;62(10):364-74. PMID 15683091
- [Background] Weatherall DJ. The inherited diseases of hemoglobin are an emerging global health burden. Blood. 2010 Jun 3;115(22):4331-6. doi: 10.1182/blood-2010-01-251348. Epub 2010 Mar 16. PMID 20233970
- [Background] Hassell KL. Population estimates of sickle cell disease in the U.S. Am J Prev Med. 2010 Apr;38(4 Suppl):S512-21. doi: 10.1016/j.amepre.2009.12.022. PMID 20331952
- [Background] Grosse SD, Odame I, Atrash HK, Amendah DD, Piel FB, Williams TN. Sickle cell disease in Africa: a neglected cause of early childhood mortality. Am J Prev Med. 2011 Dec;41(6 Suppl 4):S398-405. doi: 10.1016/j.amepre.2011.09.013. PMID 22099364
- [Background] Odievre MH, Verger E, Silva-Pinto AC, Elion J. Pathophysiological insights in sickle cell disease. Indian J Med Res. 2011 Oct;134(4):532-7. PMID 22089617
- [Background] Kanter J, Kruse-Jarres R. Management of sickle cell disease from childhood through adulthood. Blood Rev. 2013 Nov;27(6):279-87. doi: 10.1016/j.blre.2013.09.001. Epub 2013 Sep 19. PMID 24094945
- [Background] Quinn CT, Rogers ZR, McCavit TL, Buchanan GR. Improved survival of children and adolescents with sickle cell disease. Blood. 2010 Apr 29;115(17):3447-52. doi: 10.1182/blood-2009-07-233700. Epub 2010 Mar 1. PMID 20194891
- [Derived] Conde M, Lespessailles E, Wanneveich M, Allemandou D, Boulain T, Dimitrov G. Effect of nutritional supplementation on bone mineral density in children with sickle cell disease: protocol for an open-label, randomised controlled clinical trial. BMJ Open. 2024 Apr 5;14(4):e080235. doi: 10.1136/bmjopen-2023-080235. PMID 38580373